CLINICAL TRIAL: NCT03125564
Title: A Randomised, Placebo-controlled Study on Fecal Microbiota Transplantation for Patients With Irritable Bowel Syndrome With Fecal and Mucosal Microbiota Assessment
Brief Title: FMT for Patients With IBS With Fecal and Mucosal Microbiota Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMT-IBS study
Record Dates: First submitted 2017-04-07; First posted 2017-04-24 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Irritable Bowel Syndrome; Fecal Microbiota Transplantation
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Fecal Microbiota Transplantation; salicylhydroxamic acid; Defecation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal Microbiota Transplantation (Experimental): FMT infusion and Fecal and Mucosal Microbiota Assessment
  Interventions: Procedure: Fecal Microbiota Transplantation; Procedure: Fecal and Mucosal Microbiota Assessment
- Sham infusion (Sham Comparator): Infusion with sham and Fecal and Mucosal Microbiota Assessment
  Interventions: Procedure: Sham; Procedure: Fecal and Mucosal Microbiota Assessment

INTERVENTIONS:
Procedure: Fecal Microbiota Transplantation — Fecal microbiota transplantation
  Arms: Fecal Microbiota Transplantation
Procedure: Sham — Infusion of sham
  Arms: Sham infusion
Procedure: Fecal and Mucosal Microbiota Assessment — To assess the fecal and mucosal microbiota before and after Fecal Microbiota Transplantation

SUMMARY:
Irritable bowel syndrome (IBS) is a common functional bowel disorder of the gastrointestinal tract affecting up to 20 percent of the adolescent and adult populations. It is characterised by abdominal pain, irregular bowel habits, altered stool consistencies and bloating, and is associated with impaired quality of life. IBS can be categorised into diarrhoea predominant type (IBS-D), constipation predominant type (IBS-C), and mixed type (IBS-M). Fecal microbiota transplantation (FMT) defined as infusion of feces from healthy donors to affected subjects has shown impressive results with high cure rates in patients with recurrent clostridium difficile infections. The investigators propose a randomised, placebo-controlled trial of FMT in patients with IBS.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a common functional bowel disorder of the gastrointestinal tract affecting up to 20 percent of the adolescent and adult populations. It is characterised by abdominal pain, irregular bowel habits, altered stool consistencies and bloating, and is associated with impaired quality of life. IBS can be categorised into diarrhoea predominant type (IBS-D), constipation predominant type (IBS-C), and mixed type (IBS-M). Until recently, the development of an effective therapy for this condition has been hampered by a poor understanding of the etiology of the disease. Traditionally the underlying pathogenesis of IBS has been centered on the brain-gut axis whereby stress and psychological conditions alter the perception of IBS symptoms. Emerging evidence however supports the observation that at least in a subgroup of patients with IBS, peripheral mechanisms within the intestine including low grade mucosal inflammation, abnormal immune activation and altered visceral sensitivity may be the main drivers of the manifestations in IBS.

Accumulating data suggest that the intestinal microbiota play an important role in the pathophysiology of IBS. This is derived from early observation that post-infectious IBS developed in a subgroup of patients following a bout of gastroenteritis. Several studies have shown that the fecal microbiota was altered in IBS and IBS symptoms can be improved by therapeutic interventions that target the microbiota including antibiotics, probiotics and prebiotics. Rifaximin, an oral, non-systemic broad spectrum antibiotics has also been shown to provide significant relief in IBS symptoms in a randomized controlled trial.

Fecal microbiota transplantation (FMT) defined as infusion of feces from healthy donors to affected subjects has shown impressive results with high cure rates in patients with recurrent clostridium difficile infections.The mechanism of FMT in IBS is not completely clear.

The investigators propose a randomised, placebo-controlled trial of FMT in patients with IBS.

ELIGIBILITY:
Inclusion Criteria:

* Patients are aged 18 or above
* Patients have a diagnosis of IBS consistent with the Rome III criteria (13)
* Patients did not have adequate relief of global IBS symptoms and of IBS-related bloating at both the time of screening and the time of randomization
* Patients had undergone clinical investigations with colonoscopy within five years of recruitment
* Patients with written informed consent form provided

Exclusion Criteria:

* Patients have constipation predominant IBS (according to the definition of Rome III criteria)
* Patients have a history of inflammatory bowel disease or gastrointestinal malignancy
* Patients have previous abdominal surgery (other than cholecystectomy or appendectomy)
* Patients have human immunodeficiency virus infection
* Patients have renal disease manifested by 1.5 times the ULN of serum creatinine or blood urea nitrogen level
* Patients have hepatic disease manifested by twice the upper limit of normal (ULN) for any of the following liver function tests: alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, or total bilirubin (except in isolated elevation of unconjugated bilirubin
* Patients have diabetes mellitus manifested by HbA1C > 6.5%
* Patients have abnormal thyroid function manifested by values of serum Sensitive Thyroid Stimulating Hormone and serum free T4 fall outside the reference range which is not controlled by thyroid medications
* Patients have a history of psychiatric illness (mania and schizophrenia)
* Patients have depression defined by having a Patient Health Questionnaire-9 (PHQ-9) score > 15
* Patients have anxiety defined by having a Generalized Anxiety Disorder 7 (GAD7) score > 10
* Patients have active infection at the time of inclusion
* Patients have used antibiotic therapy or anti-inflammatory drugs within the past 7 days
* Patients have any other organic causes that can explain the symptoms of IBS
* Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2023-12-16 (Actual)

PRIMARY OUTCOMES:
the proportion of responders | 12 weeks
  Response means a symptom relief of more than 50 points assessed by IBS-SSS.

SECONDARY OUTCOMES:
The proportion of patients who had adequate relief of general IBS symptoms | 12 weeks
  Adequate relief of general IBS symptoms
Assess the onset and duration of relief of general IBS symptoms | 12 weeks
  The onset and duration of relief of general IBS symptoms
The proportion of patients who had improvement on abdominal bloating | 12 weeks
  Proportion of patients who had improvement on abdominal bloating between the treatment arms.
Assess the onset and duration of abdominal bloating relief | 12 weeks
  The onset and duration of abdominal bloating relief were assessed by phone interview and follow-up visits.
Assess the Abdominal pain between two groups | 12 weeks
  Assess abdominal pain by symptoms diary between treatment and placebo arms. The symptoms diary assesses abdominal pain on a scale of 0-10 and higher scores mean severe abdominal pain
Assess the Stool consistency between two groups | 12 weeks
  Assess stool consistency by Bristol Stool Scale between treatment and placebo arms. The Bristol Stool Scale ranges from 1 to 7.
Health-related quality of life in patients with irritable bowel syndrome | 12 weeks
  Assess quality of life by Irritable Bowel Syndrome Quality of Life (IBS-QOL) scale between treatment and placebo arms. The IBS-QOL scale ranges from 0 to 100 scores with higher scores indicating better quality of life.
Assess the level of anxiety between two groups | 12 weeks
  Assess the Anxiety scale by General Anxiety Disorder-7 (GAD-7) between treatment and placebo arms. The total scores of GAD-7 range from 0 to 21 with higher scores indicating more severe level of anxiety.
Assess the change of abdominal pain scores in patients who undergo open-label FMT | 12 weeks
  After unblinding, patients in the placebo group will be given a choice to receive open-label FMT and follow up under the same schedule as the blinded phase. The abdominal pain scores will be assessed by symptoms diary on a scale of 0-10 and higher scores mean severe abdominal pain
The proportion of patients who undergo open-label FMT and have abdominal bloating relief | 12 weeks
  After unblinding, patients in the placebo group will be given a choice to receive open-label FMT and follow up under the same schedule as the blinded phase. The abdominal bloating relief was assessed by phone interview and follow-up visits.
The IBS quality of life change in patients who undergo open-label FMT | 12 weeks
  After unblinding, patients in the placebo group will be given a choice to receive open-label FMT and follow up under the same schedule as the blinded phase. Quality of life was assessed by Irritable Bowel Syndrome Quality of Life (IBS-QOL) scale which ranges from 0 to 100 scores with higher scores indicating better quality of life.
The level of anxiety change in patients who undergo open-label FMT | 12 weeks
  After unblinding, patients in the placebo group will be given a choice to receive open-label FMT and follow up under the same schedule as the blinded phase. Anxiety was assessed by General Anxiety Disorder-7 (GAD-7). The total scores of GAD-7 range from 0 to 21 with higher scores indicating more severe level of anxiety.
The changes in diversity and richness of gut microbiota | 12 weeks
  Evaluating the changes in the diversity (shannon index) and richness (number of observed species) of gut microbiota of patients receiving FMT or placebo
The changes in gut microbiota at species and functional levels | 12 weeks
  Assessing changes in gut microbiota at species and functional levels in patients receiving FMT or placebo
The similarity of gut microbiota to donors | 12 weeks
  Assessing the similarity of gut microbiota to donors in patients following FMT

CONTACTS AND LOCATIONS:
Overall Officials: Siew Ng, Prof., Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilson S, Roberts L, Roalfe A, Bridge P, Singh S. Prevalence of irritable bowel syndrome: a community survey. Br J Gen Pract. 2004 Jul;54(504):495-502. PMID 15239910
- [Background] Talley NJ, Spiller R. Irritable bowel syndrome: a little understood organic bowel disease? Lancet. 2002 Aug 17;360(9332):555-64. doi: 10.1016/S0140-6736(02)09712-X. PMID 12241674
- [Background] Collins SM. A role for the gut microbiota in IBS. Nat Rev Gastroenterol Hepatol. 2014 Aug;11(8):497-505. doi: 10.1038/nrgastro.2014.40. Epub 2014 Apr 22. PMID 24751910
- [Background] Kassinen A, Krogius-Kurikka L, Makivuokko H, Rinttila T, Paulin L, Corander J, Malinen E, Apajalahti J, Palva A. The fecal microbiota of irritable bowel syndrome patients differs significantly from that of healthy subjects. Gastroenterology. 2007 Jul;133(1):24-33. doi: 10.1053/j.gastro.2007.04.005. Epub 2007 Apr 14. PMID 17631127
- [Background] Ng SC, Lam EF, Lam TT, Chan Y, Law W, Tse PC, Kamm MA, Sung JJ, Chan FK, Wu JC. Effect of probiotic bacteria on the intestinal microbiota in irritable bowel syndrome. J Gastroenterol Hepatol. 2013 Oct;28(10):1624-31. doi: 10.1111/jgh.12306. PMID 23800182
- [Background] Gwee KA, Graham JC, McKendrick MW, Collins SM, Marshall JS, Walters SJ, Read NW. Psychometric scores and persistence of irritable bowel after infectious diarrhoea. Lancet. 1996 Jan 20;347(8995):150-3. doi: 10.1016/s0140-6736(96)90341-4. PMID 8544549
- [Background] Spiller R, Campbell E. Post-infectious irritable bowel syndrome. Curr Opin Gastroenterol. 2006 Jan;22(1):13-7. doi: 10.1097/01.mog.0000194792.36466.5c. PMID 16319671
- [Background] Parkes GC, Sanderson JD, Whelan K. Treating irritable bowel syndrome with probiotics: the evidence. Proc Nutr Soc. 2010 May;69(2):187-94. doi: 10.1017/S002966511000011X. Epub 2010 Mar 18. PMID 20236566
- [Background] Pimentel M, Lembo A, Chey WD, Zakko S, Ringel Y, Yu J, Mareya SM, Shaw AL, Bortey E, Forbes WP; TARGET Study Group. Rifaximin therapy for patients with irritable bowel syndrome without constipation. N Engl J Med. 2011 Jan 6;364(1):22-32. doi: 10.1056/NEJMoa1004409. PMID 21208106
- [Background] van Nood E, Dijkgraaf MG, Keller JJ. Duodenal infusion of feces for recurrent Clostridium difficile. N Engl J Med. 2013 May 30;368(22):2145. doi: 10.1056/NEJMc1303919. No abstract available. PMID 23718168
- [Derived] Yau YK, Su Q, Xu Z, Tang W, Ching JYL, Mak JWY, Cheung CP, Fung M, Ip M, Chan PKS, Wu JCY, Chan FKL, Ng SC. Randomised clinical trial: Faecal microbiota transplantation for irritable bowel syndrome with diarrhoea. Aliment Pharmacol Ther. 2023 Oct;58(8):795-804. doi: 10.1111/apt.17703. Epub 2023 Sep 5. PMID 37667968